CLINICAL TRIAL: NCT02454062
Title: A Phase I, Open-Label, Non-Randomized, Dose-Escalating Safety, Tolerability and Pharmacokinetic Study of TAS-114 in Combination With S-1 in Patients With Advanced Solid Tumors
Brief Title: A Trial of TAS-114 in Combination With S-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-114-102; 2012-002674-31 (EudraCT Number)
Record Dates: First submitted 2015-05-11; First posted 2015-05-27 (Estimated); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors
Keywords: Phase I; Solid Tumors; Pharmacokinetics; Pharmacodynamics; MTD
MeSH Terms: interventions — TAS-114; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation TAS-114 (PART 1) (Experimental): Each cycle will be 21 days: 14 days of treatment and 7 days recovery. TAS-114 and S-1 will be escalated according to a defined dosing table and specific DLT criteria.
  Interventions: Drug: TAS-114; Drug: S-1
- Expansion phase TAS-114 (PART 2) (Experimental): The TAS-114 and S-1 MTD established in the Dose Escalation Phase will be administered BID for 14 days followed by a 7 day recovery period.
  This regimen is repeated every 21 days thereafter. Approximately 40 to 60 evaluable patients will be enrolled in the Expansion Phase. PGx, PD and PK analysis will be performed based on specific criteria.
  Interventions: Drug: TAS-114; Drug: S-1

INTERVENTIONS:
Drug: TAS-114 — TAS-114 is an inhibitor of dUTPase, a gatekeeper protein in pyrimidine-metabolism.
Drug: S-1 — S-1 is an oral antimetabolite; a combination of three pharmacological compounds: tegafur (FT), gimeracil (CDHP), and oteracil (Oxo)

SUMMARY:
A Phase I, Open-Label, International, Multicenter, Non-Randomized, Dose-Escalating Safety, Tolerance and Pharmacokinetic Study of Oral Administration of TAS-114 in Combination with S-1 in a Twice Daily Schedule for 14 Days in Patients with Advanced Solid Tumors.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, dose-escalation Phase I study of TAS-114 administered in combination with S-1, evaluating the safety, tolerability, pharmacokinetics and preliminary antitumor activity of the TAS-114/S-1 regimen in patients with advanced solid tumors.

The study will be conducted in two parts: a Dose-Escalation Phase (Part 1) to determine the MTD; and an Expansion Phase (Part 2) to further evaluate the safety and preliminary efficacy with the MTD. Patients will receive the study medication according to the proposed treatment schedule until disease progression (PD), occurrence of intolerable side effects, removal by the Investigator or withdrawal of consent. A patient is considered discontinued from study treatment when TAS-114 is discontinued.

Male or female patients age 18 years or older with confirmed advanced solid tumor(s) for which no standard therapy exists.

TAS-114/S-1 will be administered BID for 14 days followed by a 7-day recovery period, every 21 days (1 cycle) in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent.
2. Is ≥18 years of age
3. Has histologically or cytologically confirmed advanced or metastatic solid tumor(s) for which no standard therapy exists.
4. Expansion Phase only: Has at least one measurable lesion
5. Is able to take medications orally (e.g., no feeding tube).
6. Has adequate organ function
7. Women of child-bearing potential must have a negative pregnancy test (urine or serum) within 7 days prior to starting the study drug.
8. Is willing and able to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Has received treatment with any proscribed treatments within specified time frames prior to study drug administration.
2. Has a serious illness or medical condition(s)
3. Is receiving concomitant treatment with drugs that may interact with S-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12-27 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Identify Maximum Tolerated Dose (MTD) in mg/kg | Up to 2.5 Years
  To investigate the safety and determine the maximum tolerated dose (MTD) of TAS-114 in combination with S-1 in patients with advanced solid tumor(s) for which no standard therapy exists.

CONTACTS AND LOCATIONS:
Locations (5):
- Erasme University Hospital-ULB, Brussels, Belgium
- Institut Gustave Roussy, Villejuif, France
- Italy (2):
  - IRCCS San Marino IST, Genoa
  - Universita Vita-Salute San Raffaele, Milan
- IOSI Istituto Oncologico della Svizzera Italiana, Bellinzona, Switzerland

REFERENCES:
- [Background] HEIDELBERGER C, CHAUDHURI NK, DANNEBERG P, MOOREN D, GRIESBACH L, DUSCHINSKY R, SCHNITZER RJ, PLEVEN E, SCHEINER J. Fluorinated pyrimidines, a new class of tumour-inhibitory compounds. Nature. 1957 Mar 30;179(4561):663-6. doi: 10.1038/179663a0. No abstract available. PMID 13418758
- [Background] Longley DB, Harkin DP, Johnston PG. 5-fluorouracil: mechanisms of action and clinical strategies. Nat Rev Cancer. 2003 May;3(5):330-8. doi: 10.1038/nrc1074. PMID 12724731
- [Background] Shirasaka T. Development history and concept of an oral anticancer agent S-1 (TS-1): its clinical usefulness and future vistas. Jpn J Clin Oncol. 2009 Jan;39(1):2-15. doi: 10.1093/jjco/hyn127. Epub 2008 Dec 3. PMID 19052037
- [Background] Peters GJ, Backus HH, Freemantle S, van Triest B, Codacci-Pisanelli G, van der Wilt CL, Smid K, Lunec J, Calvert AH, Marsh S, McLeod HL, Bloemena E, Meijer S, Jansen G, van Groeningen CJ, Pinedo HM. Induction of thymidylate synthase as a 5-fluorouracil resistance mechanism. Biochim Biophys Acta. 2002 Jul 18;1587(2-3):194-205. doi: 10.1016/s0925-4439(02)00082-0. PMID 12084461
- [Background] Fukushima M, Satake H, Uchida J, Shimamoto Y, Kato T, Takechi T, Okabe H, Fujioka A, Nakano K, Ohshimo H, Takeda S, Shirasaka T. Preclinical antitumor efficacy of S-1: a new oral formulation of 5-fluorouracil on human tumor xenografts. Int J Oncol. 1998 Oct;13(4):693-8. doi: 10.3892/ijo.13.4.693. PMID 9735397
- [Background] Shirasaka T, Shimamoto Y, Fukushima M. Inhibition by oxonic acid of gastrointestinal toxicity of 5-fluorouracil without loss of its antitumor activity in rats. Cancer Res. 1993 Sep 1;53(17):4004-9. PMID 7689420
- [Background] Van Cutsem E, Moiseyenko VM, Tjulandin S, Majlis A, Constenla M, Boni C, Rodrigues A, Fodor M, Chao Y, Voznyi E, Risse ML, Ajani JA; V325 Study Group. Phase III study of docetaxel and cisplatin plus fluorouracil compared with cisplatin and fluorouracil as first-line therapy for advanced gastric cancer: a report of the V325 Study Group. J Clin Oncol. 2006 Nov 1;24(31):4991-7. doi: 10.1200/JCO.2006.06.8429. PMID 17075117
- [Background] Johnston PG, Fisher ER, Rockette HE, Fisher B, Wolmark N, Drake JC, Chabner BA, Allegra CJ. The role of thymidylate synthase expression in prognosis and outcome of adjuvant chemotherapy in patients with rectal cancer. J Clin Oncol. 1994 Dec;12(12):2640-7. doi: 10.1200/JCO.1994.12.12.2640. PMID 7989939
- [Background] Johnston PG, Lenz HJ, Leichman CG, Danenberg KD, Allegra CJ, Danenberg PV, Leichman L. Thymidylate synthase gene and protein expression correlate and are associated with response to 5-fluorouracil in human colorectal and gastric tumors. Cancer Res. 1995 Apr 1;55(7):1407-12. PMID 7882343
- [Background] Lenz HJ, Leichman CG, Danenberg KD, Danenberg PV, Groshen S, Cohen H, Laine L, Crookes P, Silberman H, Baranda J, Garcia Y, Li J, Leichman L. Thymidylate synthase mRNA level in adenocarcinoma of the stomach: a predictor for primary tumor response and overall survival. J Clin Oncol. 1996 Jan;14(1):176-82. doi: 10.1200/JCO.1996.14.1.176. PMID 8558194
- [Background] Peters GJ, van der Wilt CL, van Groeningen CJ, Smid K, Meijer S, Pinedo HM. Thymidylate synthase inhibition after administration of fluorouracil with or without leucovorin in colon cancer patients: implications for treatment with fluorouracil. J Clin Oncol. 1994 Oct;12(10):2035-42. doi: 10.1200/JCO.1994.12.10.2035. PMID 7931471
- [Background] Aschele C, Debernardis D, Casazza S, Antonelli G, Tunesi G, Baldo C, Lionetto R, Maley F, Sobrero A. Immunohistochemical quantitation of thymidylate synthase expression in colorectal cancer metastases predicts for clinical outcome to fluorouracil-based chemotherapy. J Clin Oncol. 1999 Jun;17(6):1760-70. doi: 10.1200/JCO.1999.17.6.1760. PMID 10561213
- [Background] Ichikawa W, Takahashi T, Suto K, Yamashita T, Nihei Z, Shirota Y, Shimizu M, Sasaki Y, Hirayama R. Thymidylate synthase predictive power is overcome by irinotecan combination therapy with S-1 for gastric cancer. Br J Cancer. 2004 Oct 4;91(7):1245-50. doi: 10.1038/sj.bjc.6602139. PMID 15354215
- [Background] Ladner RD. The role of dUTPase and uracil-DNA repair in cancer chemotherapy. Curr Protein Pept Sci. 2001 Dec;2(4):361-70. doi: 10.2174/1389203013380991. PMID 12374095
- [Background] Quesada-Soriano I, Casas-Solvas JM, Recio E, Ruiz-Perez LM, Vargas-Berenguel A, Gonzalez-Pacanowska D, Garcia-Fuentes L. Kinetic properties and specificity of trimeric Plasmodium falciparum and human dUTPases. Biochimie. 2010 Feb;92(2):178-86. doi: 10.1016/j.biochi.2009.10.008. Epub 2009 Oct 29. PMID 19879316
- [Background] Canman CE, Radany EH, Parsels LA, Davis MA, Lawrence TS, Maybaum J. Induction of resistance to fluorodeoxyuridine cytotoxicity and DNA damage in human tumor cells by expression of Escherichia coli deoxyuridinetriphosphatase. Cancer Res. 1994 May 1;54(9):2296-8. PMID 8162567
- [Background] Koehler SE, Ladner RD. Small interfering RNA-mediated suppression of dUTPase sensitizes cancer cell lines to thymidylate synthase inhibition. Mol Pharmacol. 2004 Sep;66(3):620-6. doi: 10.1124/mol.66.3.. PMID 15322254
- [Background] Ladner RD, Lynch FJ, Groshen S, Xiong YP, Sherrod A, Caradonna SJ, Stoehlmacher J, Lenz HJ. dUTP nucleotidohydrolase isoform expression in normal and neoplastic tissues: association with survival and response to 5-fluorouracil in colorectal cancer. Cancer Res. 2000 Jul 1;60(13):3493-503. PMID 10910061
- [Background] Nobili S, Napoli C, Landini I, Morganti M, Cianchi F, Valanzano R, Tonelli F, Cortesini C, Mazzei T, Mini E. Identification of potential pharmacogenomic markers of clinical efficacy of 5-fluorouracil in colorectal cancer. Int J Cancer. 2011 Apr 15;128(8):1935-45. doi: 10.1002/ijc.25514. PMID 20560137
- [Background] Takatori H, Yamashita T, Honda M, Nishino R, Arai K, Yamashita T, Takamura H, Ohta T, Zen Y, Kaneko S. dUTP pyrophosphatase expression correlates with a poor prognosis in hepatocellular carcinoma. Liver Int. 2010 Mar;30(3):438-46. doi: 10.1111/j.1478-3231.2009.02177.x. Epub 2009 Nov 30. PMID 19968781
- [Background] McIntosh EM, Haynes RH. dUTP pyrophosphatase as a potential target for chemotherapeutic drug development. Acta Biochim Pol. 1997;44(2):159-71. PMID 9360704
- [Background] Wilson PM, Fazzone W, LaBonte MJ, Deng J, Neamati N, Ladner RD. Novel opportunities for thymidylate metabolism as a therapeutic target. Mol Cancer Ther. 2008 Sep;7(9):3029-37. doi: 10.1158/1535-7163.MCT-08-0280. PMID 18790783
- [Background] Hayashi T, Yamaguchi S, Kito S, Tanaka G, Kurokawa K, Hirota T. [An oral repeated dose toxicity study of a new antineoplastic agent S-1 in dogs. I. A 13-week repeated dose toxicity study. II. An ophthalmologic toxicity recovery study]. J Toxicol Sci. 1996 Nov;21 Suppl 3:527-44. doi: 10.2131/jts.21.supplementiii_527. Japanese. PMID 9021660
- [Background] Zhu AX, Clark JW, Ryan DP, Meyerhardt JA, Enzinger PC, Earle CC, Fuchs CS, Regan E, Anbe H, Houghton M, Zhang J, Urrea P, Kulke MH. Phase I and pharmacokinetic study of S-1 administered for 14 days in a 21-day cycle in patients with advanced upper gastrointestinal cancer. Cancer Chemother Pharmacol. 2007 Feb;59(3):285-93. doi: 10.1007/s00280-006-0265-y. Epub 2006 Jun 20. PMID 16786333
- [Background] Benson AB 3rd, Ajani JA, Catalano RB, Engelking C, Kornblau SM, Martenson JA Jr, McCallum R, Mitchell EP, O'Dorisio TM, Vokes EE, Wadler S. Recommended guidelines for the treatment of cancer treatment-induced diarrhea. J Clin Oncol. 2004 Jul 15;22(14):2918-26. doi: 10.1200/JCO.2004.04.132. PMID 15254061
- [Background] American Society of Clinical Oncology; Kris MG, Hesketh PJ, Somerfield MR, Feyer P, Clark-Snow R, Koeller JM, Morrow GR, Chinnery LW, Chesney MJ, Gralla RJ, Grunberg SM. American Society of Clinical Oncology guideline for antiemetics in oncology: update 2006. J Clin Oncol. 2006 Jun 20;24(18):2932-47. doi: 10.1200/JCO.2006.06.9591. Epub 2006 May 22. PMID 16717289
- [Background] Du Bois D, Du Bois EF. A formula to estimate the approximate surface area if height and weight be known. 1916. Nutrition. 1989 Sep-Oct;5(5):303-11; discussion 312-3. No abstract available. PMID 2520314
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Saito K, Nagashima H, Noguchi K, Yoshisue K, Yokogawa T, Matsushima E, Tahara T, Takagi S. First-in-human, phase I dose-escalation study of single and multiple doses of a first-in-class enhancer of fluoropyrimidines, a dUTPase inhibitor (TAS-114) in healthy male volunteers. Cancer Chemother Pharmacol. 2014 Mar;73(3):577-83. doi: 10.1007/s00280-014-2383-2. Epub 2014 Jan 23. PMID 24452393
- [Background] Ajani JA, Rodriguez W, Bodoky G, Moiseyenko V, Lichinitser M, Gorbunova V, Vynnychenko I, Garin A, Lang I, Falcon S. Multicenter phase III comparison of cisplatin/S-1 with cisplatin/infusional fluorouracil in advanced gastric or gastroesophageal adenocarcinoma study: the FLAGS trial. J Clin Oncol. 2010 Mar 20;28(9):1547-53. doi: 10.1200/JCO.2009.25.4706. Epub 2010 Feb 16. PMID 20159816